CLINICAL TRIAL: NCT04971707
Title: Individualized Exercise Training Based on the Heart Rate Variability in Coronary Heart Disease Patient
Acronym: HRV-Predict
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Principal Investigator, Louis Bherer, Associate scientific director, Direction of prevention, Montreal Heart Institute, Montreal Heart Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2021-2897
Record Dates: First submitted 2021-07-12; First posted 2021-07-21 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Diseases; Cardiac rehabilitation; exercise training; heart rate variability; cognitive performance
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: parallel assignment, 2 groups (1:1)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This clinical trial is a double-blinded study. Patients, and research personnel performing the outcome assessments and investigators will be blinded to group allocation. Only the kinesiologists will be aware of the group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard exercise training (Active Comparator): The physical exercises intervention will include a standardized aerobic exercises training, three sessions per week for 3 months.
  Interventions: Other: Standardized exercise training
- HRV-guided exercise training (Experimental): The physical exercises intervention will include an individualized aerobic exercises training, three sessions per week for 3 months.
  Interventions: Other: HRV-guided exercise training

INTERVENTIONS:
Other: Standardized exercise training — HRV index will be measured every morning during 5 min. This group will benefit from the standard cardiovascular rehabilitation program combining both continuous moderate exercise sessions (MICT) and high intensity interval exercise sessions (HIIT). MICT sessions will be performed 2 times per week and HIIT sessions will be performed once a week.
  Arms: standard exercise training
Other: HRV-guided exercise training — HRV index will be measured every morning during 5 min. This group will benefit from the individualized cardiovascular rehabilitation program. Daily exercise (MICT, HIIT, or active recovery) will be prescribed according to the HRV-index measured on the morning of the session.
  Arms: HRV-guided exercise training

SUMMARY:
The objective of this project is to assess the effectiveness of a new modality of prescribing the intensity of physical exercise in cardiovascular rehabilitation programs according to physiological criteria (heart rate variability measured every morning) in comparison to a standard non-individualized program.

DETAILED DESCRIPTION:
In coronary artery disease patients, cardiovascular rehabilitation (CR) reduces cardiac mortality by 30% when compared to usual drug therapy without CR. Cardiorespiratory fitness (VO2peak) is the most powerful independent prognostic marker of longevity. An improvement in VO2peak is also associated with better cognitive performance in the elderly.

The effectiveness of CR varies between patients. About 25% of coronary disease patients do not improve their VO2peak after taking part of a CR program. The risk of acute event for those "non-responder" patients, (i.e. not increasing their VO2peak), is high with a mortality rate three times higher compared to "responder" individuals.

It seems that the autonomic nervous system (ANS) is playing an important role in exercise training-induced physiological responses. Based on this, it has been proposed in healthy subjects to prescribe each exercise session according to ANS parameters (via heart rate variability, HRV). It has been suggested that high-intensity exercise when HRV parameters are stable, results in better adaptations to training. Conversely, recovery sessions when HRV is impaired seem necessary.

44 participants with stable coronary artery diseases, and taking part in a CR program will be included in this study. All participants will have signed a written consent form before taking part in the study. Patients will be randomly assigned to one of the 2 following study arms: 1/ standard exercise training ; 2/ Heart Rate Variability-guided exercise training.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease patient from the Montreal Heart Institute
* Age> 18 years old
* Referred to the EPIC center in a cardiovascular rehabilitation program due to stable angina pectoris, acute coronary syndrome (with or without ST segment elevation) or after complete coronary revascularization (primary or elective) by Percutaneous Coronary Intervention.
* Able to perform a maximal cardiopulmonary exercise stress test in accordance with current cardiovascular rehabilitation recommendations.
* Able to read, understand and sign the information and consent form.

Exclusion Criteria:

* Any absolute and relative contraindication to the maximal exercise test and / or physical activity.
* Recent cardiovascular events (cardiac decompensation or treatment with positive inotropic drugs or angioplasty less than 10 days, cardiac surgery less than 1 month, valve disease requiring surgical correction, active myopericarditis, severe ventricular arrhythmias not stabilized under treatment).
* Revascularization by coronary artery bypass grafting
* Atrial fibrillation
* Renal failure
* Heart failure
* Diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Change in cardiorespiratory fitness | Baseline and post-intervention at 3 months
  Maximum incremental cardiopulmonary exercise test (VO2 max (ml.kg.min))
Responders and non-responders proportion | Baseline and post-intervention at 3 months
  Proportion in each group (%) Responders will be defined as an increased of 5% of VO2max.

SECONDARY OUTCOMES:
Parasympathetic activity | Baseline and post-intervention at 3 months
  Root Mean Square of the Successive Differences ( RMSSD) of heart rate variability (ms)
Parasympathetic activity | Baseline and post-intervention at 3 months
  High Frequency power ( HF) of heart rate variability (ms2)
heart rate variability | Baseline and post-intervention at 3 months
  Global heart rate variability : standard deviation of the normal sinus beats (SDNN, ms)
Baroreflex gain | Baseline and post-intervention at 3 months
  Baroreflex sensibility (ms/mmHg)
Change in general cognitive functioning | Baseline and post-intervention at 3 months
  Montreal Cognitive Assessment (0-30 score, with a higher score indicating a better cognitive functioning).
Change in processing speed | Baseline and post-intervention at 3 months
  Validated remote version of neuropsychological tests and iPad tests (Composite Z-score).
Change in executive functions | Baseline and post-intervention at 3 months
  Validated remote version of neuropsychological tests and iPad tests (Composite Z-score).
Change in episodic memory | Baseline and post-intervention at 3 months
  Validated remote version of neuropsychological tests (Composite Z-score).

OTHER OUTCOMES:
Change in anxiety | Baseline and post-intervention at 3 months
  State-Trait Anxiety Inventory questionnaire (Score ranges from 20-80, with a higher score indicating higher anxiety).
Change in depressive symptoms | Baseline and post-intervention at 3 months
  Geriatric Depression Scale questionnaire (Score ranges from 0-30, with a higher score indicating larger depressive symptomatology).
Change in sleep quality | Baseline and post-intervention at 3 months
  Pittsburgh Sleep Quality Index questionnaire (Score ranges from 0-21, with a higher score indicating worse sleep quality). symptomatology). symptomatology).

CONTACTS AND LOCATIONS:
Overall Officials: Louis Bherer, PhD, Principal Investigator — Montreal Heart Institute
Locations (1):
- Preventive medicine and physical activity centre (centre EPIC), Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No